CLINICAL TRIAL: NCT05301270
Title: The Effect of Dynamic Postural Changes on Muscle Activation, Kinematic Parameters and Investigation of Balance Strategies in Transtibial and Transfemoral Amputees
Brief Title: The Dynamic Postural Changes in Transtibial and Transfemoral Amputees
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mustafa Cem TÜRKMEN, Principal Investigator, Hacettepe University
Other Study IDs: GO 21/1105
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Amputation; EMG; Balance; Perturbation
Keywords: Transtibial amputee; Transfemoral amputee; EMG; Balance; Perturbation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Transtibial Amputees: Individuals aged 18-45 years, with unilateral transtibial amputation, traumatic amputation cause, using prosthesis for at least 1 year, no skin lesions-open wound on the stump, no phantom sensation or pain, no musculoskeletal problems that may affect balance other than amputation will be included.
  Interventions: Diagnostic Test: EMG Evaluation
- Transfemoral Amputees: Individuals aged 18-45 years, with unilateral transfemoral amputation, traumatic amputation cause, using prosthesis for at least 1 year, no skin lesions-open wound on the stump, no phantom sensation or pain, no musculoskeletal problems that may affect balance other than amputation will be included.
  Interventions: Diagnostic Test: EMG Evaluation
- Healthy Subjects: Healthy individuals between the ages of 18-45 will be included.
  Interventions: Diagnostic Test: EMG Evaluation

INTERVENTIONS:
Diagnostic Test: EMG Evaluation — Muscle activations in the lower extremity and trunk muscles during compensatory postural responses will be evaluated. The Delsys Trigno IM (Delsys Inc. Natick, Massachusetts, USA) wireless surface electromyography (EMG) system will be used to evaluate muscle activation. In the lower extremity; Muscle activations of tibialis anterior, gastrocnemius, quadriceps and hamstring muscle groups and erector spinae in the trunk will be evaluated. While the muscle groups above the stump on the amputated side of the individuals in the amputation group will be evaluated, all muscle groups specified on the healthy side will be evaluated. In the control group, all muscle groups on the dominant side, but on the non-dominant side, all other muscles except the tibialis anterior and gastrocnemius muscles will be evaluated in order to be compatible with the amputation group.
  Other Names: Balance Assessment; Analysis Method with Video Recording

SUMMARY:
This research was planned to examine how unpredictable movements on the support surface will affect muscle activation and kinematic parameters in individuals with transtibial and transfemoral amputations. Individuals aged between 18-45 years, using prostheses for at least 1 year, able to stand and walk independently without a walking aid, and volunteered to participate in the study with unilateral transtibial and unilateral transfemoral amputation, and healthy individuals similar to these individuals in terms of age and gender will be included in the study.

DETAILED DESCRIPTION:
This research was planned to examine how unpredictable movements on the support surface will affect muscle activation and kinematic parameters in individuals with transtibial and transfemoral amputations. Individuals aged between 18-45 years, using prostheses for at least 1 year, able to stand and walk independently without a walking aid, and volunteered to participate in the study with unilateral transtibial and unilateral transfemoral amputation, and healthy individuals similar to these individuals in terms of age and gender will be included in the study. The number of cases considered to be included in the study will be determined by the number of individuals required for the power of the study to be 0.80 in the interim statistical analysis to be made after including 5 individuals, since no similar studies on the subject could be found. After determining the number of individuals to be included in the study group, a control group consisting of the same number of healthy individuals will be formed. The amount of body weight on the intact leg and prosthetic limb of individuals with amputation "L.A.S.A.R." with the posture device, artificial limb (prosthesis) awareness will be evaluated with the "Forgotten Joint Score-12" scale. Posture assessment of all individuals will be carried out by photogrammetric method. Dynamic balance evaluations of all participants will be made with the "Bertec balance device". Afterwards, the compensatory postural responses of all individuals, which are formed by the movements of the platform in the sagittal plane at an unpredictable moment, while standing on the motor-assisted and controllable movable platform, will be evaluated. Muscle activations occurring in both lower extremity and trunk muscles during compensatory postural responses will be evaluated with the "Delsys Trigno IM wireless surface electromyography (sEMG) system". Simultaneously, the motion will be recorded with the camera from the sagittal plane and the "Dartfish Analysis Software" software will be used for the analysis of the video images obtained. By using video recording and analysis method, angular changes in the joints during body oscillations, segment positions and balance strategies used will be examined. As a result of our research, it is anticipated to determine whether there is a difference between transtibial, transfemoral amputation and healthy individuals in terms of balance strategies resulting from unexpected surface perturbations, muscle activations in the lower extremities and trunk, and kinematic changes. In addition, it is anticipated to determine whether there is a relationship between dynamic balance values and lower extremity and trunk muscle activations that occur with unexpected surface perturbations in transtibial amputated, transfemoral amputated and healthy individuals. Thus, it is thought that the biomechanical properties of compensatory postural responses, which are very important in terms of maintaining postural control in individuals with transtibial amputation and transfemoral amputation, will contribute to the current scientific knowledge.

ELIGIBILITY:
Inclusion Criteria:

For all groups;

* After giving detailed information about the research, those who volunteered to participate in the research
* Able to stand and walk independently without any walking aid
* They are determined as individuals with cooperation who can understand tests and evaluations.

For Amputation Groups;

* Having unilateral transtibial or transfemoral amputation,
* The cause of amputation is traumatic,
* Functional classification is at the level of K2 and K3 (Medicare Functional Classification Level),
* Using prosthesis for at least 1 year,
* No skin lesion or open wound on the stump,
* No phantom sensation or pain
* It was determined as individuals who do not have musculoskeletal problems (muscle shortness, limitation of joint movement, etc.) that may affect balance other than amputation.

Exclusion Criteria:

For all groups;

* Known orthopedic (except amputation for the amputee group), neurological disease, vestibular problems, severe visual impairment, cognitive dysfunction,
* Having pain originating from the musculoskeletal system (Also for the amputation group; stump pain or the presence of pain caused by the use of prosthesis),
* Individuals who exercise regularly,
* With a history of serious trauma,
* History of falling in the last 1 year,
* Pain during measurement of maximal voluntary contraction,
* It was determined as individuals with a body mass index (BMI)>30 kg/m².

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with amputation to be included in the study (study group); It will consist of individuals who agree to participate in the research with transtibial or transfemoral amputation followed at Hacettepe University Faculty of Physical Therapy and Rehabilitation, Prosthesis and Biomechanics Unit and Bilim Orthotics Prosthesis Application Center.
  The control group, on the other hand, will consist of volunteers from patients' relatives and employees at Hacettepe University Faculty of Physical Therapy and Rehabilitation and Bilim Orthotics Prosthesis Application Center, who are similar to the study group in terms of age and gender.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Muscle activations | Day 0
  Evaluation of muscle activations of lower extremity and trunk muscles with sEMG
Percent Maximum Voluntary İsometric Contraction (MVIC) | Day 0
  In order to normalize the muscles whose activations will be evaluated as percent MVIC, MVIC values will be measured in muscle test positions, which are the positions where the muscles are most activated.
Analysis with video recording | Day 0
  Data obtained by video recording on individuals on a platform that can move in the sagittal plane will be obtained and analyzed with Dartfish software.
Balance Assessment | Day 0
  Dynamic balance assessment will be performed with the Bertec BalanceCheck Screener™ BP5050 20x20 inc device (Bertec BP5050 balance plate platform; Bertec, Corp., Columbus, OH, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Semra Topuz, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No